CLINICAL TRIAL: NCT06778889
Title: Assessing the Impacts of Physical Activity on Mental Health and Perceived Stress Among Undergraduate Medical Students in Pakistan: a Cross-Sectional Study
Brief Title: Assessing the Impacts of Physical Activity on Mental Health and Perceived Stress Among Undergraduate Medical Students in Pakistan
Status: Completed | Type: Observational
Sponsor: Rawalpindi Medical College (Other)
Responsible Party: Principal Investigator, Nazeer Ahmed, Final year medical student, Rawalpindi Medical College
Other Study IDs: KMDC-PA-MH-2025
Record Dates: First submitted 2025-01-03; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Mental Health; Perceived Stress; Physical Activity
Keywords: Mental Health profile; Perceived Stress; Medical students; Physical activity
MeSH Terms: conditions — Psychological Well-Being; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Undergraduate Medical Students: This cohort consists of undergraduate medical students enrolled in the medical program. They will be assessed for their physical activity levels, perceived stress, and mental health.
  Interventions: Behavioral: Undergraduate Medical Students

INTERVENTIONS:
Behavioral: Undergraduate Medical Students — This is an observational study without any intervention. Data will be collected using standardized questionnaires to assess physical activity, mental health, and stress levels in the participants.

SUMMARY:
Brief Summary

The goal of this observational study is to understand how physical activity affects mental health and perceived stress in undergraduate medical students in Pakistan. The main questions it aims to answer are:

Does physical activity improve the mental health of medical students? Does physical activity lower the stress levels of medical students?

Researchers will compare students who engage in physical activity to those who do not to see if physical activity improves their mental health and reduces stress.

Participants will:

Complete surveys about their mental health and perceived stress. Report their physical activity levels, including how often they exercise and for how long.

This study will help identify how lifestyle changes, like exercising, can improve the well-being of medical students and potentially reduce the challenges they face during their education.

DETAILED DESCRIPTION:
Detailed Description

This observational, cross-sectional study investigates the relationship between physical activity and its effects on mental health and perceived stress among undergraduate medical students in Pakistan. The study aims to determine whether engaging in regular physical activity can improve psychological well-being and reduce perceived stress in this population, which is known to face significant academic and personal stressors during their medical education.

Study Objectives and Rationale

Medical students encounter a variety of stressors, including demanding coursework, clinical responsibilities, and personal challenges. This study aims to provide a quantitative assessment of how physical activity can mitigate these stressors and improve mental health outcomes. It hypothesizes that students engaging in higher levels of physical activity will exhibit better mental health and lower perceived stress.

Study Design and Methodology

Study Design:

Observational, cross-sectional study. Data collected at a single time point using validated self-reported questionnaires.

Study Setting:

The study was conducted in both public and private medical colleges across Pakistan, providing a diverse sample of participants.

Data Collection Tools:

International Physical Activity Questionnaire (IPAQ-7): Used to measure physical activity levels, categorized as low, moderate, or high based on MET-minutes per week. Perceived Stress Scale (PSS-10): Used to quantify perceived stress levels. Scores are categorized as low (0-13), moderate (14-26), and high (27-40). Brief Symptom Inventory (BSI-18): Measures psychological distress, including somatization, depression, and anxiety, with a composite Global Severity Index (GSI).

Data Collection Procedure:

Participants were invited to complete online surveys distributed via Google Forms. Data collected included demographic information, physical activity habits (frequency, intensity, duration), stress levels, and mental health status. All participants provided informed consent, and confidentiality was maintained throughout the study.

Data Analysis Plan:

Descriptive statistics: Used to summarize participant demographics, activity levels, and mental health profiles. Inferential statistics: Chi-square tests to assess associations between physical activity levels and stress/mental health outcomes. Regression analysis to examine the predictive role of physical activity on mental health and perceived stress, adjusting for confounding factors such as age, gender, and academic year.

Study Duration:

The study was conducted over six months, with data collection completed within this timeframe. Key Technical Considerations The IPAQ-7 questionnaire quantifies physical activity in MET-minutes per week, allowing categorization into low (<600 MET-minutes/week), moderate (600-3000 MET-minutes/week), and high (>3000 MET-minutes/week) activity levels. The BSI-18 generates individual scores for somatization, depression, and anxiety, and calculates a composite GSI score (range: 0-72), where higher scores indicate greater psychological distress. Statistical analysis will control for potential confounders, ensuring robust interpretation of results. Significance and Potential Impact

This study will provide evidence on how physical activity can improve mental health and reduce stress among medical students in Pakistan, a population particularly vulnerable to mental health challenges. Findings may inform the development of interventions and institutional policies that integrate physical activity into student support systems to promote psychological well-being and academic success.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate medical students from any academic year.
* Students who are willing to participate and provide informed consent.
* Students who engage in physical activity (any frequency or duration) within the last month

Exclusion Criteria:

* Students who do not provide informed consent.
* Students with physical disabilities or medical conditions that prevent participation in physical activity (e.g., severe cardiovascular conditions, musculoskeletal disorders).
* Students with a diagnosed mental health disorder that may interfere with the study's focus on stress and mental health (e.g., schizophrenia, bipolar disorder).
* Students with language barriers.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will target undergraduate medical students aged 18-30 years from various institutions. The population will include both male and female students, ensuring a comprehensive analysis of mental health, perceived stress, and physical activity.
Sampling Method: Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Mental Health Status of Undergraduate Medical Students | Data have been collected once during the survey period, which spans from February 2 to October 2, 2024.
  The primary outcome measure is to assess the mental health status of undergraduate medical students using the Brief Symptom Inventory-18 (BSI-18), which assesses psychological distress across three subscales: anxiety, depression, and somatization. The BSI-18 uses a 5-point Likert scale, where 0 = "not at all" and 4 = "extremely," to measure each symptom's intensity.
  The Global Severity Index (GSI) is calculated from the total score across all subscales, with higher scores indicating higher distress. The subscale scores for anxiety, depression, and somatization range from 0 to 24, where higher scores reflect greater psychological discomfort.
  Minimum value: 0 (indicating no distress)Maximum value: 24 (indicating extreme distress)
  In addition to raw scores, the BSI-18 also provides T-scores (mean = 50, SD = 10) for each subscale, allowing for comparison across populations regardless of their distribution. Higher T-scores indicate more significant distress.

SECONDARY OUTCOMES:
Perceived Stress Levels among Undergraduate Medical Students. | Data have been collected once during the survey period, which spans from February 2 to October 2, 2024.
  The secondary outcome measure is to assess the perceived stress levels of undergraduate medical students using the Perceived Stress Scale (PSS-10), which assesses perceived stress over the past month. The PSS-10 includes 10 items rated on a 5-point scale (0 = "never" to 4 = "very often"). The total score ranges from a minimum value of 0 (indicating no perceived stress) to a maximum value of 40 (indicating very high perceived stress). Higher scores represent worse outcomes, reflecting greater levels of perceived stress. The interpretation is as follows:
  Low stress: 0-13 Moderate stress: 14-26 High stress: 27-40

OTHER OUTCOMES:
Physical Activity Levels of Undergraduate Medical Students | Data have been collected once during the survey period, which spans from February 2 to October 2, 2024.
  It assess physical activity levels among undergraduate medical students using the International Physical Activity Questionnaire-7 (IPAQ-7). This will allow the study to explore the correlation between physical activity and both perceived stress and mental health.
  The IPAQ-7 measures physical activity levels based on three types of activities: walking, moderate intensity, and vigorous intensity. The total score is calculated in MET-minutes/week. Range of scores is as follows:
  Minimum value: 0 MET-minutes/week (indicating no physical activity) Maximum value: There is no upper limit; however, higher values reflect higher physical activity levels.
  Higher scores indicate better outcomes, representing higher levels of physical activity, which are generally associated with better mental health and lower perceived stress. The physical activity levels are categorized as:
  Low activity: 0-599 MET-minutes/weekModerate activity: 600-2999 MET-minutes/weekHigh activity: 3000+ MET-minutes/week

CONTACTS AND LOCATIONS:
Overall Officials: Nazeer Ahmed, MBBS, Principal Investigator — Karachi medical and dental college karachi Pakistan
Locations (1):
- Karachi medical and dental college, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that support the findings of this study will be shared, including data related to mental health profiles, perceived stress levels, and physical activity levels obtained from BSI-18, PSS-10, and IPAQ-7 questionnaires.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The IPD and supporting information will be available starting 6 months after publication and will remain accessible for 5 years.
Access Criteria: Researchers who provide a methodologically sound proposal to investigate questions relevant to the study objectives will have access. Proposals should be directed nazeermed313@gmail.com. Data will be made available through a secure online repository after approval.

REFERENCES:
- Available data/document: Study Protocol — https://orcid.org/0009-0009-6142-6201 — Data and supporting documents, including the study protocol, statistical analysis plan, and anonymized data set, will be available upon request to the corresponding author (email: nazeermed313@gmail.com) starting [insert date]. Requests will be reviewed based on a valid research purpose and agreement to use data ethically